CLINICAL TRIAL: NCT01142271
Title: Comparison of Billroth-I and Roux-en-Y Reconstruction After Distal Subtotal Gastrectomy for Gastric Cancer Patients : Prospective Randomized Study
Brief Title: Comparison of Billroth-I and Roux-en-Y Reconstruction After Distal Subtotal Gastrectomy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, Sang-Uk Han, Department of Surgery, Ajou University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AJIRB-MED-DEO-09-297
Record Dates: First submitted 2010-06-08; First posted 2010-06-11 (Estimated); Last update posted 2011-11-07 (Estimated); Status verified 2011-11

CONDITIONS: Gastrectomy
Keywords: Distal gastrectomy; Reconstruction; Reflux; subtotal gastrectomy
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Gastroenterostomy; Anastomosis, Roux-en-Y; Gastric Bypass

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Billroth-I (Experimental): Patients in this group should be underwent gastroduodenostomy as reconstruction procedure after standard distal subtotal gastrectomy with lymph node dissection.
  Interventions: Procedure: Billroth-I
- Roux en Y (Experimental): Patients in this group should be underwent jejunojejunostomy and gastrojejunostomy as reconstruction procedure after standard distal gastrectomy.
  Interventions: Procedure: Roux en Y

INTERVENTIONS:
Procedure: Billroth-I — Standard distal gastrectomy with D1 plus beta or D2 lymph node dissection would be performed for distal gastric cancer. After that, gastroduodenostomy should be performed by circular stapler. In addition, stapler sites were re-enforced.
  Other Names: Gastroduodenostomy
  Arms: Billroth-I
Procedure: Roux en Y — Standard distal gastrectomy with D1 plus beta or D2 lymph node dissection would be performed for distal gastric cancer. After that, jejunojejunostomy and gastrojejunostomy should be performed by circular staplers. In addition, stapler sites were re-enforced.
  Other Names: Gastrojejunostomy and jejunojejunostomy
  Arms: Roux en Y

SUMMARY:
The purpose of this trial is to compare the degree of reflux, operative outcomes and quality of life between Roux en Y and Billroth-I reconstructions after distal subtotal gastrectomy for gastric cancer

DETAILED DESCRIPTION:
Most common procedure for the resection of gastric cancers located in middle or lower stomach is distal subtotal gastrectomy. However, the optimal reconstruction procedure after that has still not to be established. Although B-I reconstruction is most common method due to the safety and simplicity, the duodenal fluid may reflux into the remnant stomach which may contribute to the mucosal injury to remnant stomach and esophagus. Roux en Y reconstruction may reduce the reflux to remnant stomach due to the length of Roux en Y limb, although it is more complicated procedure.

Therefore, we plan to collect 120 patients to compare the degree of reflux between Roux en Y and Billroth-I reconstructions after distal subtotal gastrectomy for gastric cancer. In addition, we compare the surgical outcome and quality of life between two groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with adenocarcinoma at the endoscopic biopsy
* Patients who are possible to be performed curative resection in imaging study
* Patients with tumor which not involved in pylorus and are located in mid or distal portion of the stomach
* Patients with informed consent
* Patients with three or less American Society Anesthesiology Score 3

Exclusion Criteria:

* Patients who are or become pregnant
* Patients with uncontrolled disease
* Patient s with synchronous other malignancy
* Patients participated in other clinical trial

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2010-06; Primary Completion 2012-05 (Estimated); Study Completion 2012-05 (Estimated)

PRIMARY OUTCOMES:
Reflux of bile content | 6 months after surgery
  We estimate the degree of reflux by gastrofiberscopic findings using reflux score suggested by Romaganoli. In addition, histological finding of remnant stomach by endoscopic biopsy is also investigated. Reflux symptom is surveyed by Gastrointestinal Symptom Rating Scale.

SECONDARY OUTCOMES:
Quality of Life | 6 months after surgery
  We investigate the quality of life with EORTC-C30, EORTC-STO22 questionnaire suggested by European Organization for Research and Treatment of Cancer (EORTC).
Morbidity | 2 month after surgery
  We investigate the occurrence of complication during recovery after surgery.
Anastomotic time | Day 1
  We estimate anastomosis time
Nutritional state | 6 month after surgery
  We estimate Albumin, transferrin, lymphocyte, body weight
Mortality | 2 month after operation
  We investigate the occurrence of operation-related death during recovery after surgery.
Operation time | Day 1
  We estimate total operation time.

CONTACTS AND LOCATIONS:
Overall Officials: Sang-Uk Han, M.D., Ph D., Principal Investigator — Department of Surgery, Ajou University School of Medicine; Hoon Hur, M.D., Study Director — Department of Surgery, Ajou University School of Medicine
Locations (1):
- Ajou University Hospital, Suwon, South Korea

REFERENCES:
- [Background] Chan DC, Fan YM, Lin CK, Chen CJ, Chen CY, Chao YC. Roux-en-Y reconstruction after distal gastrectomy to reduce enterogastric reflux and Helicobacter pylori infection. J Gastrointest Surg. 2007 Dec;11(12):1732-40. doi: 10.1007/s11605-007-0302-0. Epub 2007 Sep 18. PMID 17876675
- [Background] Ishikawa M, Kitayama J, Kaizaki S, Nakayama H, Ishigami H, Fujii S, Suzuki H, Inoue T, Sako A, Asakage M, Yamashita H, Hatono K, Nagawa H. Prospective randomized trial comparing Billroth I and Roux-en-Y procedures after distal gastrectomy for gastric carcinoma. World J Surg. 2005 Nov;29(11):1415-20; discussion 1421. doi: 10.1007/s00268-005-7830-0. PMID 16240061
- [Derived] Nishizaki D, Ganeko R, Hoshino N, Hida K, Obama K, Furukawa TA, Sakai Y, Watanabe N. Roux-en-Y versus Billroth-I reconstruction after distal gastrectomy for gastric cancer. Cochrane Database Syst Rev. 2021 Sep 15;9(9):CD012998. doi: 10.1002/14651858.CD012998.pub2. PMID 34523717
- [Derived] Hur H, Ahn CW, Byun CS, Shin HJ, Kim YB, Son SY, Han SU. A Novel Roux-en-Y Reconstruction Involving the Use of Two Circular Staplers after Distal Subtotal Gastrectomy for Gastric Cancer. J Gastric Cancer. 2017 Sep;17(3):255-266. doi: 10.5230/jgc.2017.17.e32. Epub 2017 Sep 26. PMID 28970956